CLINICAL TRIAL: NCT04483453
Title: Effect of Nutritional Intervention on Metabolic Response in Infants: A Single-Blind, Randomized, Controlled Trial
Brief Title: Effect of Nutritional Intervention on Metabolic Response in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18.17.INF
Record Dates: First submitted 2020-07-06; First posted 2020-07-23 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Infant Development; Glucose, High Blood

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXPL feeding regimen (Experimental): Lower protein / lower estimated glycemic index regimen
  Interventions: Other: EXPL feeding regimen
- CTRL feeding regimen (Active Comparator): Standard protein / standard glycemic index regimen
  Interventions: Other: CTRL feeding regimen

INTERVENTIONS:
Other: EXPL feeding regimen — EXPL FUF (lower protein and 100% lactose) + EXPL IC (whole grains and legumes)
  Arms: EXPL feeding regimen
Other: CTRL feeding regimen — CTRL FUF (standard protein content and carbohydrate profile) + CTRL IC (refined grains)
  Arms: CTRL feeding regimen

SUMMARY:
The purpose of this study is to determine the glucose response of complementary feeding regimens consisting of two different follow-up formulas (FUFs) and infant cereals (ICs).

DETAILED DESCRIPTION:
This is a prospective, randomized, single-blind, controlled, 2-arm parallel group trial in infants aged 6 months (26 weeks) at enrollment, who are no longer breastfed, and who are ready but have not yet started complementary feeding. They will be fed one of two different isocaloric feeding regimens (Experimental [EXPL] or Control [CTRL]) consisting of different follow-up formulas (FUFs) and infant cereals (ICs). The main purpose of this study is to determine the glucose response of these two different complementary feeding regimens. All enrolled infants will participate in the trial for approximately 6 months.

ELIGIBILITY:
Inclusion Criteria:.

1. Written informed consent has been obtained from both parent / liable parent or legally acceptable representative (LAR), if applicable
2. Healthy infant who was singleton, full-term gestational birth (≥ 37 completed weeks of gestation) with a birth weight of ≥ 2.5 kg and ≤ 4.5 kg
3. Infant is no longer breastfeeding or receiving breast milk, has not yet started FUF, and is developmentally ready to begin complementary feeding
4. Infant's parent(s)/guardian is of legal age of consent, must understand the informed consent form and other study documents, and is willing and able to fulfill the requirements of the study protocol.
5. At screening visit (visit 0), infant is 24 - 26 weeks (5½ - 6 months) old
6. Weight-for-height value >-2 standard deviations from the WHO Child Growth Standards median

Exclusion Criteria:

1. Chronic infectious, metabolic, or other disease including any condition that in the opinion of the investigator may impact feeding, growth or adherence to study procedures
2. Major congenital or chromosomal abnormality known to affect growth (e.g., congenital heart disease, cystic fibrosis)
3. Known or suspected cows' milk protein intolerance / allergy, or lactose intolerance, gluten sensitivity or severe food allergies that impact diet
4. Born to mothers with gestational diabetes or type 1 diabetes
5. Major medical/surgical event requiring prolonged hospitalization during the first 6 months
6. Receiving or having received insulin, growth hormone or any other medication known to affect glucose or carbohydrate metabolism or pre- or probiotics known to affect fecal microbiota prior to enrollment
7. Subjects or subjects' parent(s) or legal representative who are not willing and not able to comply with scheduled visits and the requirements of the study protocol
8. Currently participating or having participated in another clinical trial within 4 weeks prior to trial start

Ages: 24 Weeks to 26 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2020-07-31 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Glucose peak | Study days 85-92
  Average of the glucose peaks measured by a continuous glucose monitor

SECONDARY OUTCOMES:
Glycemic response | Study days 85-92
  Incremental area under the blood glucose response curve
Glucose response variability | Study days 85-92
  Mean amplitude of glycemic excursions, standard deviation, J-index
Skinfold thickness | age 6 months, 9 months, and 12 months
  Subscapular and triceps skinfold thicknesses
Weight | age 6 months, 9 months, and 12 months
  Weight (g)
Length | age 6 months, 9 months, and 12 months
  Length (cm)
Head circumference | age 6 months, 9 months, and 12 months
  Head circumference (cm)
Body mass index (BMI) | age 6 months, 9 months, and 12 months
  Weight and height will be combined to report BMI in kg/m^2
Weight-for-age z-score | age 6 months, 9 months, and 12 months
  Weight-for-age z-score based on World Health Organization (WHO) growth charts
Weight-for-length z-score | age 6 months, 9 months, and 12 months
  Weight-for-length z-score based on WHO growth charts
Length-for-age z-score | age 6 months, 9 months, and 12 months
  Length-for-age z-score based on WHO growth charts
Head circumference-for-age z-score | age 6 months, 9 months, and 12 months
  Head circumference-for-age z-score based on WHO growth charts
BMI-for-age z-score | age 6 months, 9 months, and 12 months
  BMI-for-age z-score based on WHO growth charts
Insulin secretion | age 6 months, 9 months, and 12 months
  Urinary C-peptide:creatinine ratio
Dietary intake | age 6 months, 9 months, and 12 months
  Total energy, carbohydrate and protein intake calculated from food recalls / diaries
Stool microbiota composition | age 6 months, 7.5 months, 9 months, and 12 months
  Fecal microbiota composition assessed using next generation sequencing
Stool pH | age 6 months, 7.5 months, 9 months, and 12 months
  Stool pH
Stool microbiota metabolism | age 6 months, 7.5 months, 9 months, and 12 months
  Stool organic acids
Gastrointestinal (GI) tolerance | age 6 months, 9 months, and 12 months
  GI tolerance assessed using the Infant Gastrointestinal Symptom Questionnaire (IGSQ). IGSQ scores range from 13 to 65, with lower scores indicating lower GI symptom burden.
Health-related quality of life | age 6 months, 9 months, and 12 months
  Health-related quality of life using the Infant and Toddler Quality of Life Questionnaire Short Form (ITQOL-SF47). ITQOL-SF47 scores range from 0 to 100, with higher scores indicating a more favorable health-related quality of life.

OTHER OUTCOMES:
Insulin-like growth factor-1 (IGF-1) | age 6 months, 9 months, and 12 months
  Urinary IGF-1
Urinary metabolomic profile | age 6 months, 9 months, and 12 months
  Untargeted analysis of urine metabolites by H1-nuclear magnetic resonance (NMR) spectroscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Las Piñas Doctors Hospital, Las Piñas, Philippines

IPD SHARING:
Plan to Share IPD: Undecided